CLINICAL TRIAL: NCT01993251
Title: Does Melatonin Restore Sleep Architecture in Autistic Children?
Brief Title: Does Melatonin Restore Sleep Architecture in Autistic Children
Acronym: SOMELIA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-732; 2013-001230-17 (EudraCT Number)
Record Dates: First submitted 2013-11-13; First posted 2013-11-25 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Sleep Disorders
Keywords: sleep,melatonin,autism,children
MeSH Terms: conditions — Sleep Wake Disorders | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- melatonin 0.5mg (Active Comparator)
  Interventions: Drug: melatonin
- melatonin 2mg (Active Comparator)
  Interventions: Drug: Melatonin
- melatonin 6mg (Active Comparator)
  Interventions: Drug: Melatonin
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: melatonin — one capsule, melatonin 0.5 mg, oral, once a day, 30 minutes before bedtime
  Arms: melatonin 0.5mg
Drug: Melatonin — one capsule, melatonin 2 mg, oral, once a day, 30 minutes before bedtime
  Arms: melatonin 2mg
Drug: Melatonin — one capsule, melatonin 6 mg, oral, once a day, 30 minutes before bedtime
  Arms: melatonin 6mg
Drug: placebo — one capsule, placebo, oral, once a day, 30 minutes before bedtime
  Arms: placebo

SUMMARY:
Although behavioral disorders origins in autistic children are still unclear, they seem to be influenced by sleep disorders. Results of studies performed on sleep quality in autistic children showed a high prevalence of sleep disorders in these children, estimated between 50 and 80% compared to children with typical development and insomnia is one of the sleep disorders most frequently reported by autistic children's parents. Others studies showed circadian rhythm disorder in autistic children which could be the consequence of genetic abnormalities in the melatonin synthesis and the melatonin role in the synaptic transmission modulation.

Melatonin by its sedative effects and its action on circadian pacemaker is a promoter of sleep proposed for insomnia treatment and circadian rhythm disorders.

Two major recent studies (not yet published) in the United States and in England seek to show the effectiveness of melatonin by testing the effects of three doses of melatonin on reducing sleep disorders.

It is therefore interesting and important to conduct a parallel study to assess the melatonin effect not only on the reduction of sleep disorders (sleep onset latency, total sleep time…), but on sleep quality (number of nocturnal awakenings).

The strength of this study lies in the combination of several measurement tools to assess the melatonin dose-effect on all parameters in both physiological (actimetrics, polysomnography), biological (dosage 24h sulfatoxymelatonin), behavioral (sleep questionnaire, index of insomnia severity, rating scale autistic disorder) as well as possible side effects.

The primary objective is to determine the most effective dose of melatonin to improve sleep quality in autistic children.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls from 3 to 12 years old with autism spectrum,
* Diagnosed by psychiatrists according to the diagnostic criteria for autism ICD-10 AND ADI or ADOS positive,
* With trouble sleeping, assessed by questionnaire CHSQ,
* Having made a night polysomnography,
* Written informed consent (signed by parents),
* Affiliated with the French universal healthcare system.

Exclusion Criteria:

* Children who stopped all treatment for sleep for less than one month,
* Liver or kidney insufficiencies,
* Acute illness during or occurred in the month preceding the study,
* Neurological disease without autism spectrum , patients with non-controlled epilepsy
* Health background witch can influence sleep (other than autism itself),
* Obstructive syndrome (history - oral breathing in wakefulness, nocturnal snoring significant (heard the door closed), nocturnal respiratory effort, apnea reported by parents- and clinical examination (chronic nasal congestion, large tonsils and touching),
* Known hypersensitivity to the active substance or to one of the excipient contained in the verum or in the placebo,
* Children under treatment against-indicated with the study treatment witch can't be stopped

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
To determine the most effective dose of melatonin to improve sleep quality in autistic children. | The primary outcome will be assessed once at V2 (D29 +/- 7days) by polysomnography.
  The primary outcome is to measure the awakenings index which is the number of nocturnal awakenings higher than 15 seconds per hour of sleep measured by polysomnography.

SECONDARY OUTCOMES:
To assess in autistic children the melatonin effects on sleep characteristics | It will be assessed once at V2 (D29 +/- 7 days) by polysomnography and actimetrics.
  by measuring the sleep latency
To assess the effectiveness of treatment on sleep disorders. | It will be assessed once at V2 (D29 +/- 7 days) by polysomnography and actimetrics.
  It is to evaluate the effectiveness with the scale treatment response, the sleep questionnaire and severity index of insomnia
To assess the effectiveness of melatonin on daytime autistic behavior | It will be assessed three times at V1 (D0), V2 (D29 +/- 7 days) and V4 (D44+/-7days).
  Evaluate the effectiveness with the rating scale autistic behavior.
To assess the melatonin safety in autistic children. | It will be assessed three times at V2 (D29 +/- 7 days), V3(D30) and V4 (D44+/-7days).
  Evaluate the safety with Adverse events report.
Establish whether there is a correlation between sleep quality and melatonin secretion. | It will be assessed twice at V3 (D30) and V4 (D44+/-7days).
  With the urinary melatonin dosage.
To assess in autistic children the melatonin effects on sleep characteristics. | at V2 (D29 +/- 7 days) by polysomnography and actimetrics.
  by measuring the indexes arousals
To assess in autistic children the melatonin effects on sleep characteristics. | at V2 (D29 +/- 7 days) by polysomnography and actimetrics.
  by measuring time and percentage of different stages of NREM (Non rapid eye movement) and REM sleep
To assess in autistic children the melatonin effects on sleep characteristics | at V2 (D29 +/- 7 days) by polysomnography and actimetrics
  by measuring the density of sleep spindles in light NREM sleep
To assess in autistic children the melatonin effects on sleep characteristics | at V2 (D29 +/- 7 days) by polysomnography and actimetrics.
  by measuring the density of eye movements REM sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Franco, MD, Principal Investigator — CHU Hôpital Femme Mère Enfant.Bron
Locations (5):
- France (5):
  - Hôpital Femme Mere Enfant, Bron
  - CHU de Caen, Caen
  - Centre Hospitalier du Chinonais, Chinon
  - CHRU de Strasbourg, Strasbourg
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Effects of immediate melatonin on sleep and behavior in children with autism SOMELIA study Guyon A, Comajuan M, Limousin N, Trippi, Schröder C, Plancoulaine S, Franco P The 21st International Congress of the ESCAP - Beyond nature & nurture Strasbourg, France, 29/06/2025 - 01/07/2025